CLINICAL TRIAL: NCT04645498
Title: Prospective Study on the Impact of COVID-19 on the Equilibrium of Hereditary Metabolic Disease (MHM) in Patients With or Who Have Contracted COVID-19
Brief Title: COVID-19 and Hereditary Metabolic Diseases
Acronym: COVID19-MHM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_52; 2020-A02886-33 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-11-25; First posted 2020-11-27 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Covid19; Metabolism, Inborn Errors
Keywords: COVID-19; Inherited metabolic diseases
MeSH Terms: conditions — COVID-19; Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metabolism, Inborn Errors: Patient affected by an inherited metabolic disease

SUMMARY:
No additional risk factors have been identified in patients with Inherited Metabolic Diseases (IMD) for contracting or presenting complications of COVID-19 compared to the general population. Yet, IMD patients have cell/tissue alterations that could constitute a potential direct or indirect target for the virus. We do not know the impact of this infection on patients suffering from MHM, nor the possible effect of specific treatment of MHM on the evolution of COVID-19.

This study will collect French IMD patients having or having had COVID-19 infection. The main objective is to estimate among IMD patients contracting COVID-19 the frequency of disease aggravation or metabolic decompensation.

The secondary objectives will be : a. to evaluate the incidence of COVID-19 diagnosed in a given group of IMD when the number of patients with this IMD is known (Urea Cycle Deficiency, Gaucher Disease). b. to evaluate the impact of IMD on the and severity of COVID-19 infection

ELIGIBILITY:
Inclusion Criteria:

* Child or adult patient with a diagnosis of IMD
* Symptomatic or asymptomatic patient tested positive for COVID-19 (PCR and/or serology)
* Symptomatic patient non tested but with strong clinical suspicion for COVID-19
* Patient affiliated with the health insurance

Exclusion Criteria:

* inability to receive informed information
* Persons deprived of liberty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IMD patients followed in reference centers for IMD in France. children and adult patients with MHM who have been infected with COVID-19 (tested positive or considered positive for COVID-19). Asymptomatic MHM patients tested positive for COVID 19 (contact case, for example) will also be studied.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Frequency of MHM imbalance triggered by COVID-19 | at 8 weeks
  disease aggravation or metabolic decompensation, among MHM-infected patients with COVID-19.

SECONDARY OUTCOMES:
Number of COVID-19 patients in Gaucher's disease | at 24 months
Number of COVID-19 patients in Urea Cycle Disorder | at 24 months
Severity of COVID-19 infection | at 24 months
  severity of COVID-19 infection as assessed by hospitalization; Intensive Care Unit, death

CONTACTS AND LOCATIONS:
Overall Officials: Claire Douillard, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France